CLINICAL TRIAL: NCT02365506
Title: A Double-blind, Placebo-controlled Study to Evaluate the Effect of GS-6615 on QT, Safety and Tolerability in Subjects With Long QT2 Syndrome
Brief Title: Study to Evaluate the Effect of Eleclazine on QT, Safety, and Tolerability in Participants With Long QT2 Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-394-1658
Record Dates: First submitted 2015-02-12; First posted 2015-02-19 (Estimated); Results first posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: LQT2 Syndrome
Keywords: Congenital Long QT Syndrome; LQTS; Sudden Cardiac Death
MeSH Terms: conditions — Long Qt Syndrome 2; Death, Sudden, Cardiac | interventions — eleclazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Eleclazine 24 mg + Eleclazine 48 mg + Placebo (Experimental): Participants will receive placebo to match eleclazine on Days 1 and 4, eleclazine 24 mg on Day 2 and eleclazine 48 mg on Day 3.
  Interventions: Drug: Eleclazine; Drug: Placebo
- Eleclazine 48 mg + Placebo (Experimental): Participants will receive placebo to match eleclazine on Days 1, 2 and 4, and eleclazine 48 mg on Day 3.
  Interventions: Drug: Eleclazine; Drug: Placebo
- Placebo (Placebo Comparator): Participants will receive placebo to match eleclazine on Days 1 to 4.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eleclazine — Tablets administered orally in a single dose
  Other Names: GS-6615
  Arms: Eleclazine 24 mg + Eleclazine 48 mg + Placebo; Eleclazine 48 mg + Placebo
Drug: Placebo — Placebo to match tablets administered orally in a single dose

SUMMARY:
The primary objective of the study is to evaluate the effect of oral eleclazine (formerly GS-6615) on corrected QT (QTc) interval in participants with long QT2 syndrome.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with an established diagnosis of LQT2 (by genotype testing)
* Mean (of triplicate) QTc interval ≥ 480 msec for at least four out of seven time points, determined by standard 12-lead electrocardiogram (ECG), at screening

Key Exclusion Criteria:

* Known mutations associated with long QT syndrome type 1 or long QT syndrome type 3
* Known or suspected history of seizures or epilepsy
* History of heart failure defined as New York Heart Association (NYHA) Class IV and/or known left ventricular ejection fraction (EF) ≤ 45%
* Body mass index (BMI) ≥ 36 kg/m^2 at screening
* Severe renal impairment at screening (defined as an estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m^2, using the 4 variable modification of diet in renal disease (MDRD) equation), as determined by the study center
* Abnormal liver function tests at screening, defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 x upper limit of normal (ULN), or total bilirubin > 1.5 x ULN
* An aborted cardiac arrest (ACA), implantable cardioverter-defibrillator (ICD) implantation, syncopal episode, or appropriate ICD therapy within 3 months prior to screening
* Any other condition or circumstance that in the opinion of the investigator would preclude compliance with the study protocol.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-07-20 (Actual); Primary Completion 2016-05-13 (Actual); Study Completion 2016-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (1):
- University of Rochester Medical Center/Strong Memorial Hospital, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 1 study site in the United States. The first participant was screened on 20 July 2015. The last study visit occurred on 13 June 2016.
Pre-assignment Details: 15 participants were screened.
Groups:
- Eleclazine 24 mg + Eleclazine 48 mg + Placebo: Participants received single oral dose of placebo to match eleclazine tablet on Days 1 and 4, a single oral dose of eleclazine 24 mg (4 x 6 mg) tablets on Day 2 and a single oral dose of eleclazine 48 mg (8 x 6 mg) tablets on Day 3.
- Eleclazine 48 mg + Placebo: Participants received single oral dose of placebo to match eleclazine tablet on Days 1, 2 and 4, and a single oral dose of eleclazine 48 mg (8 x 6 mg) tablets on Day 3.
- Placebo: Participants received placebo to match eleclazine tablets on Days 1 to 4.
Period: Overall Study
Arm/Group | Eleclazine 24 mg + Eleclazine 48 mg + Placebo | Eleclazine 48 mg + Placebo | Placebo
Started | 4 | 4 | 5
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 1
Not completed — Investigator's Discretion | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Eleclazine 24 mg + Eleclazine 48 mg + Placebo | Eleclazine 48 mg + Placebo | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 5 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (15.3) | 40 (13.9) | 48 (11.0) | 43 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 9
  Male | 1 | 1 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 4 | 5 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Standard 12-Lead Electrocardiogram (ECG) Daytime QT Interval Corrected For Heart Rate Using The Fridericia Formula (QTcF) (AUC0-8)/8 at Day 3: Lead V5
Description: Daytime (AUC0-8)/8 was defined as the area under the QTc curve during the 8 hours postdose, where 0 was defined as the time of dosing (i.e., T = 0) on a given day. Daytime (AUC0-8)/8 was computed by dividing AUC0-8 by the time from dosing to the 8 hour postdose time point. QTcF is corrected QT interval using Fridericia's formula.
Time Frame: Baseline (Day 1), Day 3
Population: Participants in the Full Analysis Set (included all participants who took at least 1 dose of study drug and had standard 12-lead Day 3 QT measurements recorded) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Eleclazine 24 mg + Eleclazine 48 mg + Placebo | Eleclazine 48 mg + Placebo | Placebo
Number analyzed (Participants) | 4 | 3 | 4
msec
  Baseline | 447.2 (5.32) | 468.3 (26.20) | 464.3 (20.50)
  Change at Day 3 | -5.3 (8.31) | 0.4 (15.20) | 2.1 (7.71)
Statistical Analysis 1: Comparison: Eleclazine 24 mg + Eleclazine 48 mg + Placebo vs Placebo; Test type: Superiority; p = 0.358, Mixed Models Analysis; p-value is from a mixed model with fixed effect for treatment, day, and treatment by day with baseline daytime QTcF as a covariate; Difference in LSM = -7.7, 95% CI 2-sided [-26.0 to 10.5], Standard Error of Mean 7.92 — Least Square mean (LSM) and 95% confidence interval (CI) is from a mixed model with fixed effect for treatment, day, and treatment by day with baseline daytime QTcF as a covariate
Statistical Analysis 2: Comparison: Eleclazine 48 mg + Placebo vs Placebo; Test type: Superiority; p = 0.840, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LSM = -1.7, 95% CI 2-sided [-20.0 to 16.7], Standard Error of Mean 7.96 — LSM and 95% CI are from a mixed model with fixed effect for treatment, day, and treatment by day with baseline daytime QTcF as a covariate

2. Primary Outcome: Change From Baseline in Standard 12-Lead ECG Daytime QTcF (AUC0-8)/8 at Day 3: Lead II
Description: Daytime (AUC0-8)/8 was defined as the area under the QTc curve during the 8 hours postdose, where 0 was defined as the time of dosing (i.e.,T = 0) on a given day. Daytime (AUC0-8)/8 was computed by dividing AUC0-8 by the time from dosing to the 8 hour postdose time point. QTcF is corrected QT interval using Fridericia's formula.
Time Frame: Baseline (Day 1), Day 3
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Eleclazine 24 mg + Eleclazine 48 mg + Placebo | Eleclazine 48 mg + Placebo | Placebo
Number analyzed (Participants) | 4 | 3 | 4
msec
  Baseline | 447.7 (5.48) | 464.7 (34.00) | 461.2 (20.01)
  Change at Day 3 | -3.4 (7.72) | 8.7 (8.96) | 3.3 (7.19)
Statistical Analysis 1: Comparison: Eleclazine 24 mg + Eleclazine 48 mg + Placebo vs Placebo; Test type: Superiority; p = 0.338, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LSM = -6.0, 95% CI 2-sided [-19.8 to 7.8], Standard Error of Mean 5.83 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Eleclazine 48 mg + Placebo vs Placebo; Test type: Superiority; p = 0.425, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LSM = 5.3, 95% CI 2-sided [-9.4 to 19.9], Standard Error of Mean 6.21 — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: Change From Baseline in Standard 12-Lead ECG Daytime QTcF (AUC0-8)/8 at Day 3: Global Lead
Description: as for outcome 1
Time Frame: Baseline (Day 1), Day 3
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Eleclazine 24 mg + Eleclazine 48 mg + Placebo | Eleclazine 48 mg + Placebo | Placebo
Number analyzed (Participants) | 4 | 4 | 4
msec
  Baseline | 453.3 (8.11) | 471.2 (41.88) | 477.9 (32.80)
  Change at Day 3 | -7.8 (7.55) | 0.5 (9.68) | -3.5 (3.90)
Statistical Analysis 1: Comparison: Eleclazine 24 mg + Eleclazine 48 mg + Placebo vs Placebo; Test type: Superiority; p = 0.174, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LSM = -6.5, 95% CI 2-sided [-16.5 to 3.5], Standard Error of Mean 4.42 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Eleclazine 48 mg + Placebo vs Placebo; Test type: Superiority; p = 0.448, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LSM = 3.4, 95% CI 2-sided [-6.3 to 13.1], Standard Error of Mean 4.28 — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Change From Baseline in Holter Daily QTcF Interval (Daytime and Nocturnal) at Day 3 : Lead V5
Description: Daily Holter QTcF interval was calculated as the average of the daytime QTcF interval (AUC0-6)/6 and nocturnal QTcF interval (AUC0-6)/6. Daytime AUC0-6 was defined as the area under the QTc curve during the 6 hours postdose and nocturnal AUC0-6 was defined as the area under the QTc curve from midnight to 6am. (AUC0-6)/6 was computed by dividing AUC0-6 by the time difference over the 6 hours. QTcF is corrected QT interval using Fridericia's formula.
Time Frame: Baseline (Day 1), Day 3
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Eleclazine 24 mg + Eleclazine 48 mg + Placebo | Eleclazine 48 mg + Placebo | Placebo
Number analyzed (Participants) | 3 | 3 | 4
msec
  Baseline | 461.6 (6.89) | 466.6 (20.00) | 481.2 (28.12)
  Change at Day 3 | 3.5 (10.37) | 7.8 (2.20) | -4.1 (13.77)
Statistical Analysis 1: Comparison: Eleclazine 24 mg + Eleclazine 48 mg + Placebo vs Placebo; Test type: Superiority; p = 0.339, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LSM = 8.8, 95% CI 2-sided [-12.0 to 29.6], Standard Error of Mean 8.50 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Eleclazine 48 mg + Placebo vs Placebo; Test type: Superiority; p = 0.178, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LSM = 12.8, 95% CI 2-sided [-7.7 to 33.4], Standard Error of Mean 8.40 — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: Change From Baseline in Holter Daily QTcF Interval (Daytime and Nocturnal) at Day 3 : Global Lead
Description: as for outcome 4
Time Frame: Baseline (Day 1), Day 3
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Eleclazine 24 mg + Eleclazine 48 mg + Placebo | Eleclazine 48 mg + Placebo | Placebo
Number analyzed (Participants) | 3 | 4 | 4
msec
  Baseline | 461.6 (7.85) | 483.3 (33.11) | 486.4 (28.03)
  Change at Day 3 | 3.2 (8.02) | 2.0 (3.81) | -0.6 (14.67)
Statistical Analysis 1: Comparison: Eleclazine 24 mg + Eleclazine 48 mg + Placebo vs Placebo; Test type: Superiority; p = 0.564, Mixed Models Analysis; Difference in LSM = 4.9, 95% CI 2-sided [-14.1 to 23.9], Standard Error of Mean 8.03
Statistical Analysis 2: Comparison: Eleclazine 48 mg + Placebo vs Placebo; Test type: Superiority; p = 0.721, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LSM = 2.7, 95% CI 2-sided [-14.7 to 20.2], Standard Error of Mean 7.38 — [estimate comment as in outcome 1, analysis 2]

6. Secondary Outcome: Maximum Reduction From Predose in Standard 12-Lead QTcF on Days 2 and 3: Lead V5
Description: Maximal reduction from predose (0 hour) is the maximum decrease from predose of the QTc interval (QTcF) at any time point from 1 to 8 hours postdose for Days 2 and 3. QTcF is corrected QT interval using Fridericia's formula. Predose was defined as the Day 2 predose value.
Time Frame: Predose, Days 2 and 3
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Eleclazine 24 mg + Eleclazine 48 mg + Placebo | Eleclazine 48 mg + Placebo | Placebo
Number analyzed (Participants) | 4 | 3 | 4
msec
  Predose | 450.6 (13.00) | 481.6 (33.28) | 453.9 (20.31)
  Day 2 | -14.3 (7.82) | -40.3 (20.85) | -9.4 (14.11)
  Day 3 | -16.3 (5.80) | -64.4 (75.73) | 2.8 (15.57)

7. Secondary Outcome: Maximum Reduction From Predose in Standard 12-Lead QTcF on Days 2 and 3: Lead II
Description: Maximal reduction from predose is the maximum decrease from predose of the QTc interval (QTcF) at any time point from 1 to 8 hours postdose for Days 2 and 3. QTcF is corrected QT interval using Fridericia's formula. Predose was defined as the Day 2 predose value.
Time Frame: Predose, Days 2 and 3
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Eleclazine 24 mg + Eleclazine 48 mg + Placebo | Eleclazine 48 mg + Placebo | Placebo
Number analyzed (Participants) | 4 | 3 | 4
msec
  Predose | 458.3 (11.54) | 482.1 (37.67) | 455.8 (21.61)
  Day 2 | -16.5 (9.34) | -37.1 (37.79) | -9.1 (18.40)
  Day 3 | -21.5 (6.14) | -35.8 (24.15) | -1.7 (18.06)

8. Secondary Outcome: Maximum Reduction From Predose in Standard 12-Lead QTcF on Days 2 and 3: Global Lead
Description: as for outcome 7
Time Frame: Predose, Days 2 and 3
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Eleclazine 24 mg + Eleclazine 48 mg + Placebo | Eleclazine 48 mg + Placebo | Placebo
Number analyzed (Participants) | 4 | 4 | 4
msec
  Predose | 458.8 (14.60) | 473.5 (42.27) | 461.7 (24.49)
  Day 2 | -18.3 (8.31) | -13.5 (6.92) | -4.6 (17.12)
  Day 3 | -23.3 (6.10) | -15.7 (14.01) | 2.1 (11.29)

ADVERSE EVENTS:
Time Frame: First dose date up to 30 days after last dose of study drug (up to Day 34)
Description: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Arm/Group | Eleclazine 24 mg + Eleclazine 48 mg + Placebo | Eleclazine 48 mg + Placebo | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 1/4 | 2/4 | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eleclazine 24 mg + Eleclazine 48 mg + Placebo (N=4) | Eleclazine 48 mg + Placebo (N=4) | Placebo (N=5)
Palpitations (Cardiac disorders) | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 3
Migraine with aura (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or The study has been completed at all study sites for at least 2 years